CLINICAL TRIAL: NCT03602092
Title: The Observational Registry: Nationwide Data Collection on Gastrointestinal Stromal Tumors (GISTs) Patients (Taiwan GISTs Registry)
Brief Title: Observational Registry Data on GIST Patients
Status: Recruiting | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government); National Taiwan University Hospital (Other); China Medical University Hospital (Other); Changhua Christian Hospital (Other); Chang Gung Memorial Hospital (Other); National Cheng-Kung University Hospital (Other); Kaohsiung Medical University (Other); Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: T1218
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Biospecimen Retention: Samples With DNA — C-KIT
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — This is a longitudinal, multi-center, registry study, collecting data via a web-based portal in patients with GIST (Gastrointestinal Stromal Tumor) from hospitals in Taiwan.

SUMMARY:
This is a longitudinal, multi-center, registry study, collecting data via a web-based portal in patients with GIST (Gastrointestinal Stromal Tumor) from hospitals in Taiwan.

DETAILED DESCRIPTION:
Research question and objectives:

This study is to collect and describe real-world data for Taiwanese GIST on:

* Prevalence and demographic characteristics of Taiwanese GIST
* Treatment pattern of GIST therapies
* Bio-marker and/or gene expression characteristics of Taiwanese GIST
* Treatment outcome of TKI therapies, including recurrence-free, progression-free and overall survival
* Safety profile for TKI therapies

Study design: Retrospective and prospective observational cohort study Population: Taiwan GIST patients during 01 January 2010 to 31 December 2020 Data sources: Medical records and investigator-established data bank Study size: Data from up to 3,000 eligible subjects will be collected Data analysis: Descriptive statistics for longitudinally assess nationwide trends on current and evolving diagnostic, treatment, and outcome measures in the GIST population and estimate the prevalence of GIST in Taiwan.

Milestones: Interim report before 31 December 2018 and final study report before 30 June 2026.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with Gastrointestinal Stromal Tumor
2. ≥20 years old
3. Histology-confirmed GIST between 01 January 2010 and 31 December 2020.
4. Patient with prospective data collection: Willing to provide singed inform-consent as per local regulatory requirements.

Exclusion Criteria:

1. Inability and unwillingness to give informed consent if required by site ethic committee.
2. Patient that is unlikely candidate to obtain long-term follow-up information for reasons of unavailability or with severe concomitant illnesses per investigator judgement

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Gastrointestinal Stromal Tumor
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-10-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To establish the database for GIST | From date of registration to 31 December 2025
  By register the clinical presentation, diagnostic, stage, treatment and clinical outcome of GIST patients.

CONTACTS AND LOCATIONS:
Overall Officials: Tsang-Wu Liu, M.D, Study Director — Taiwan Cooperation Organization Group,NHRI,Taiwan
Locations (1):
- Yu wei-lan, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No